CLINICAL TRIAL: NCT00278551
Title: Immune Ablation and Hematopoietic Stem Cell Support in Patients With Rheumatoid Arthritis and High Risk Factors
Brief Title: Stem Cell Support in Patients With Rheumatoid Arthritis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Richard Burt, MD (Other)
Responsible Party: Sponsor-Investigator, Richard Burt, MD, MD, Northwestern University
Organization: Northwestern University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 96RA1; NCT00017615 (obsolete NCT alias)
Record Dates: First submitted 2006-01-15; First posted 2006-01-18 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: RHEUMATOID ARTHRITIS
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- heatopoietic stem cell transplant (Experimental)
  Interventions: Biological: Immune ablation and hematopoietic stem cell transplant

INTERVENTIONS:
Biological: Immune ablation and hematopoietic stem cell transplant — Autologous Hematopoietic Stem Cell Transplant

SUMMARY:
Rheumatoid arthritis (RA) is a chronic illness, immunologically mediated, probably induced by the exposure to an antigen or antigens, to which immunologic tolerance is lost. The disease has a variable course, from a mild, intermittently symptomatic illness requiring only symptomatic therapy to a fulminant illness requiring dangerous immunosuppressive therapy, surgery or both. The molecular defect causing RA has not been characterized, but may involve aberrant T cell, B cell, and macrophage function. Although RA often responds to immunosuppressive medication including corticosteroids, methotrexate, azathioprine and cyclophosphamide, or to non-steroidal anti-inflammatory drugs, no therapy has been curative. In patients with severe RA, who have been unresponsive to corticosteroids, and who have more than 20 active joints or vasculitis, we propose, as a phase I-II study, complete immune ablation and subsequent reconstitution with autologous in vitro T lymphocyte depleted PBSCs harvested from the patient prior to immune ablation. The combination of high dose cyclophosphamide and anti-thymocyte globulin conditioning will be followed by rescue with autologous lymphocyte depleted PBSCs. Subsequent disease activity will be followed by: (1) RA disease activity index, (2) type and amount of therapy for RA, and (3) flow cytometry of peripheral blood lymphocyte subsets, (4) joint count, (5) patients' assessment of pain, (6) arthritis impact measurement scales (AIMS) questionnaire, (7) acute phase reactants. This study will dose standard therapy, i.e. immune suppression, to the point of complete immune ablation and subsequent recapitulation of lymphocyte ontogeny by PBSC rescue. We anticipate that this study will also form the basis to clarify further the role of the immune system in RA.

ELIGIBILITY:
Inclusion Criteria:

1. Physiologic age < 60 years old or >18 years old.
2. An established clinical diagnosis of rheumatoid arthritis by American College of Rheumatology criteria, and a positive rheumatoid factor will be required.
3. Patients must have failed two disease-modifying agents, such as methotrexate, plaquenil, gold, azathioprine, asulfidine or D-penicillamine.
4. Patients must have six (6) swollen joints from active RA and either thirty (30) or greater involved joints (swelling, tenderness, deformity, pain on motion, or decreased motion), or have answered less than 75 percent of Health Assessment Questionnaire (HAQ) questions "without any difficulty."
5. A harvest of PBSC greater than 1.4 x 106 CD34+ cells /kg after CD34+ selection will be necessary for the patient to proceed to transplant.
6. Ability to give informed consent
7. Patients with Juvenile Rheumatoid Arthritis (JRA) will be candidates if disease onset is polyarthritic or systemic and they have at least 6 swollen joints and have failed corticosteroids and two disease-modifying drugs

Exclusion Criteria:

1. HIV positive
2. History of coronary artery disease, or congestive heart failure.
3. Uncontrolled diabetes mellitus, or any other illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive chemoradiotherapy
4. Prior history of malignancy except localized basal cell or squamous skin cancer. Other malignancies for which the patient is judged to be cured by local surgical therapy, such as head and neck cancer, or stage I breast cancer will be considered on an individual basis.
5. Positive pregnancy test, inability or unwillingness to pursue effective means of birth control, failure to willingly accept or comprehend irreversible sterility as a side effect of therapy.
6. Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible
7. FEV1/FVC < 75% of predicted, DLCO < 50% of predicted.
8. Resting LVEF < 45 %
9. Bilirubin > 2.0 mg/dl, transferase (AST) > 2x upper limit of normal
10. Serum creatinine > 2.0 mg/dl
11. Platelet count less than 100,000/ul, ANC less than 1000/ul
12. History of allergy to eggs or murine proteins
13. Known hypersensitivity to E. coli derived proteins

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 1997-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Tender joint count; Swollen joint count; Patient's assessment of pain;Patient's global assessment of disease; Physician global assessment;Acute phase reactant value (erythrocyte sedimentation rate). | 5 years after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Feinberg School of Medicine, Chicago, Illinois, United States